CLINICAL TRIAL: NCT07142837
Title: A Study to Evaluate the Efficacy and Safety of ZG005 in Combination With Gecacitinib and Chemotherapy for Participants With Advanced Solid Tumors
Brief Title: Study of ZG005 in Combination With Gecacitinib and Chemotherapy for Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-JAK-004
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Dose-escalation study of ZG005 in combination with Gecacitinib and Chemotherapy.
  Interventions: Drug: ZG005; Drug: Gecacitinib
- Part 2: Dose Expansion (Experimental): Cohort A: HER2-negative gastric or gastroesophageal junction adenocarcinoma; Cohort B: Esophageal squamous cell carcinoma; Cohort C: other Solid Tumors.
  Interventions: Drug: ZG005; Drug: Gecacitinib

INTERVENTIONS:
Drug: ZG005 — ZG005 20mg/kg; once every 3 weeks；IV infusion
Drug: Gecacitinib — Gecacitinib for dose escalations are set as 100mg Bid po. Gecacitinib for dose expansion will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage.

SUMMARY:
This is a multicenter, open-label phase I/II study for participants with advanced solid tumors who have failed prior immune checkpoint inhibitor therapies.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-75 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* PART 1: Histologically confirmed unresectable locally advanced, recurrent, or metastatic solid tumors.PART 2 Cohort A: Histologically confirmed unresectable locally advanced, recurrent, or metastatic HER2-negative gastric or gastroesophageal junction adenocarcinoma. Cohort B: Histologically confirmed unresectable locally advanced, recurrent, or metastatic esophageal squamous cell carcinoma. Cohort C: Histologically confirmed unresectable locally advanced, recurrent, or metastatic other solid tumors.
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* participants were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first 28 days
Objective Response Rate (ORR) | Up to 2 years
Adverse events (AEs) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hosptial, Beijing, Beijing Municipality, China